CLINICAL TRIAL: NCT06153056
Title: Identification of Factors Predictive of the Efficacy of Endoscopic Endoscopic Sleeve Gastroplasty & Study the Evolution of Clinical, Biological and Intestinal Intestinal Microbiota After Surgery
Brief Title: Identification of Factors Predictive of the Efficacy of Endoscopic Endoscopic Sleeve Gastroplasty
Acronym: PREDISLEGE
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230882; 2023-A01226-39 (Other: IDRCB)
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Obesity
Keywords: Obesity; Endoscopic sleeve gastroplasty; Weight loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples (blood, plasmatheque, serotheque, stool) taken as part of the research will be will be collected in a biological collection. 12 mL blood on dry tube, 12 mL on EDTA tube, for a total of 24 mL of blood, will be collected at each research visit. 5 aliquots of serum and 5 aliquots of plasma of 0.5 mL will be kept. An aliquot of 1 mL of whole blood will be stored. 10 aliquots of approximately 2 mL of stool. 1 saliva swab of saliva will be collected and stored.
  These collections will be kept at the biochemistry and bacteriology laboratory of the Antoine Béclère hospital, for a period of 30 years. At the end of the research, the samples may be used for further analyses not provided for in the protocol, which may prove to be of interest. that may be of interest in the context of obesity pathology, depending on the obesity, in line with the development of scientific knowledge, subject to the patient's informed, as indicated in the information/consent form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bloed-, ontlasting- en speekselmonsters — In addition, the blood collected (24 mL) will be used for the following analyses:
  GLP-1, PYY, branched-chain amino acids, Adipokines, leptin, adiponectin Blood bile acid levels: total and detailed analyzed by HPLC MS/MS Serum microbiome profile Genome-wide association study.
  The stool sample will be used to establish the :
  Intestinal bile acid profile Intestinal microbiota profile Saliva sampling for oral microbiota profiling.

SUMMARY:
Endoscopic sleeve gastroplasty and bypass are currently available for weight loss in obese patients who have failed nutritional management. Despite very low risks, these techniques remain invasive. What's more, the French National Authority for Health recommends this procedure for patients with a BMI above 35 kg/m² with associated co-morbidities, or above 40 kg/m². This excludes grade I obese patients (30 < BMI < 35) who have no effective means of losing weight. The hospital's hepato-gastroenterology and nutrition department has therefore implemented endoscopic sleeve gastroplasty to address this problem. As with other surgical techniques, there is heterogeneity heterogeneity in weight loss. The investigators therefore aim to identify factors predictive of the efficacy of this procedure in order to improve patient management of patients.

DETAILED DESCRIPTION:
The prevalence of obesity is increasing worldwide, and it is estimated that one quarter of the world's population will be overweight or obese by 2045. Obesity can lead to complications, including cardiovascular damage (myocardial ischemia and stroke), liver damage (non-alcoholic steatohepatitis and liver cancer), diabetes and extra-hepatic cancers. In this context, achievement of a significant long-term weight loss is of paramount importance to ameliorate patient outcome. Bariatric surgery is the most effective treatment for severe obesity and results in a significant long-term weight loss. However, bariatric surgery is restricted to patients with a BMI >40 kg/m2 or >35 kg/m2 with commodities (hypertension, diabetes, sleep apnoea, NASH). Therefore, the majority of obese patients do not benefit from this procedure. Recent advances in flexible endoluminal endoscopy now provide the tools for transoral endoscopic gastric volume reduction (ESG, endoscopic sleeve gastroplasty).

The gastric body is reduced by an endoscopic procedure involving suture plications. This minimally invasive method may be a good therapeutic option to obtain a significant weight reduction in patients with moderate obesity or those with severe obesity and no indication for bariatric surgery (BMI between 35 and 40 kg/m2 without commodities). In this context this study aims to identify predictive factors of weight loss following ESG and explore changes of metabolic parameters, metabolomic profiles and gut microbiota profiles. This is a retro-prospective cohort study including patients with moderate obesity undergoing ECG between March 2017 and September 2023. Clinical parameters (weight, high, BMI, weight fluctuations), serum metabolic parameters (standard lipid profile, lipoprotein levels, fasting plasma glucose, insulin levels, C-peptide levels, hemoglobin A1c) and liver function test parameters (standard biology, transient elastometry, Fibrotest®, Actitest®, abdominal ultrasound) are systematically collected for all patients before ESG and then at three- and twelve-month post-ESG. Samples of serum, plasma, stools and saliva are also systematically collected for research purpose before ESG and then at three- and twelve-month post-ESG. Each sample is stored at -80°C for subsequent analysis. Metabolomic/lipidomic analysis will be used to quantify metabolite and lipid species in serum/plasma samples. Metagenomic analysis will be used to characterise faecal and salivary microbiota profiles.

ELIGIBILITY:
Inclusion Criteria:

* Patient of legal age (Age ≥ 18 years)
* Patient capable of understanding the study and signing a consent.
* BMI between 30 and 35 kg/m² with the presence of at least one one obesity-related complication (diabetes, dyslipidemia, sleep apnea syndrome, non-alcoholic steatohepatitis, joint pain joint pain).
* Patients with a BMI greater than 35 kg/m² who have been bariatric surgery has been refused.
* Patient who has failed to lose weight and improve with conventional techniques.
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Patient having taken antibiotics 3 months prior to inclusion.
* Patient under legal protection.
* Patient at risk of gastric cancer requiring regular endoscopic surveillance: extensive intestinal atrophy and/or metaplasia on biopsy.
* Patient with a history of gastrointestinal inflammatory disease of gastric localization, hepatic or renal insufficiency, portal hypertension.
* Patient with evidence of peptic ulcer disease and/or progressive peptic ulcer disease.
* Patient with pathology affecting general health health and/or life expectancy.
* Patient with a history of bariatric surgery.
* Patient on AME

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major grade I obese patients (BMI between 30 and 35 kg/m²) not eligible for sleeve gastrectomy
Sampling Method: Non-Probability Sample
Enrollment: 205 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2031-02-02 (Estimated); Study Completion 2031-02-02 (Estimated)

PRIMARY OUTCOMES:
Serum metabolite profile using widely targeted metabolomics according to weigh loss amount (less than 10% of total weight versus more than 10% of total weight loss at 12 months post-surgery) | Before endoscopic sleeve gastroplasty
  A volume of 50 µl of serum/plasma will be used for analysis of serum metabolites using widely targeted metabolomics mass spectrometry.

SECONDARY OUTCOMES:
Clinical parameters at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  Weight expressed in kg, percentage of total weight loss and percentage of excessed weight loss will be analysed as they are systematically available in usual clinical practice.
Basic serum lipid profile at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  Basic serum lipid profile will be analysed by spectrometry as they are systematically available in usual clinical practice.
Glycated hemoglobin at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  Glycated hemoglobin expressed in % will be analysed as they are systematically available in usual clinical practice.
Insulin at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  Insulin expressed in mUI/l will be analysed as it is systematically available in usual clinical practice.
C peptide at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  C peptide expressed in µg/l will be analysed as it is systematically available in usual clinical practice.
Ferritin at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  Ferritin expressed in µg/l will be analysed as it is systematically available in usual clinical practice.
Liver function test parameter Alanine transaminase (ALT) at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  ALT levels expressed in IU/l will be analysed as they are systematically available in usual clinical practice.
Liver function test parameter aspartate transaminase (AST) at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  AST levels expressed in IU/l will be analysed as they are systematically available in usual clinical practice.
Liver function test parameter Gamma-glutamyltransferase (GGT) at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  GGT levels expressed in IU/l will be analysed as they are systematically available in usual clinical practice.
Liver function test parameter Alkaline phosphatase (ALP) at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  ALP levels expressed in IU/l will be analysed as they are systematically available in usual clinical practice.
Liver fibrosis assessed by transient elastometry at baseline and then at 3 and 12 month post-intervention | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  Transient elastometry expressed in kPa will be analysed as they are systematically available in usual clinical practice.
Liver steatosis assessed by controlled attenuation parameter (CAP) at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  Controlled attenuation parameter expressed in dB/m will be analysed as they are systematically available in usual clinical practice.
Serum metabolites using widely targeted metabolomics at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  A volume of 50 µl of serum/plasma will be used for analysis of serum metabolites using widely targeted metabolomics by mass spectrometry
Complications of endoscopic sleeve gastroplasty | During the first week post-endoscopic sleeve gastroplasty and at Month 3 and Month 12
  Data on the potential complications (occurrence of perforation, bleeding, peritonitis and other infections, thrombo-embolic events and death) of endoscopic sleeve gastroplasty will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Cosmin VOICAN, MD, PhD, Principal Investigator — APHP, Antoine-Béclère Hospital
Locations (1):
- Hôpital Antoine Béclère, Paris, France

IPD SHARING:
Plan to Share IPD: No